CLINICAL TRIAL: NCT06439914
Title: IFN-y PET Imaging: Bench to Bedside
Brief Title: First-in-human Study of Interferon-y PET Imaging to Assess Response to Immunotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nerissa T. Viola (Other)
Responsible Party: Sponsor-Investigator, Nerissa T. Viola, Principle Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-092
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [89Zr]Zr-DFO-emapalumab (Experimental): Radiotracer [89Zr]Zr-DFO-emapalumab injection
  Interventions: Drug: [89Zr]Zr-DFO-emapalumab

INTERVENTIONS:
Drug: [89Zr]Zr-DFO-emapalumab — Radiotracer [89Zr]Zr-DFO-emapalumab administration followed by 3 PET Scans (day 0, day 1 and day 3-5) within 14 days of starting immunotherapy and repeated once 25-45 days after immunotherapy started
  Other Names: Zirconium Zr 89-DFO-emapalumab

SUMMARY:
The goal of this clinical trial is to investigate the use of [89Zr]Zr-DFO-emapalumab as an IFN-γ PET imaging agent to detect lesions and response to therapy among treatment-naïve non-small cell lung cancer (NSCLC) patients. PET scans following the imaging agent will be completed prior to and about 30 days after starting immunotherapy.

DETAILED DESCRIPTION:
Participants will be enrolled into the clinical trial once confirmed eligible. Screening activities include, standard of care blood work, medical history and a physical exam.

-Within 14 days of starting immunotherapy, participants will complete PET scans 1-2 hours post-tracer administration, again on the day following tracer administration, and 3-5 days after the tracer administration. This sequence may be repeated 25-45 days after the start of treatment with immunotherapy for a total of two tracer injections and up to six PET scans.

ELIGIBILITY:
Inclusion

* Prior histologic or cytologic diagnosis of non-small cell lung cancer.
* FDG PET done within 2 months of the baseline imaging, as part of standard-of-care.
* measurable disease by RECIST 1.1 with at least one lesion of at least 2 cm in a region of the body that can be imaged by PET (e.g.,outside of the liver)
* must be able to lie still for the tests. Their girth and weight must be suitable to enter the gantry, which varies per tomograph.
* must be >18 years old.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the cancer center.
* Physical exam, CBC and Multiphasic (including electrolytes, BUN, creatinine, total bilirubin, AST, and ALT) must be done within 28 days prior to PET imaging

Exclusion

* No prior immunotherapy for current stage of NSCLC (Non Small Cell Lung Cancer). Immunotherapy in neoadjuvant or adjuvant setting and have recurrence at least 12 months following completion of immunotherapy are eligible after discussion with the principle investigator.
* Pregnant or breast feeding individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-09-25 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
peak Standard Uptake Value (SUVpeak) | Up to Day 45
  Descriptively summarize at baseline and post-immunotherapy treatments.
mean Standard Uptake Value (SUVmean) | Up to Day 45
  Descriptively summarize at baseline and post-immunotherapy treatments.
maximum Standard Uptake Value (SUVmax) | Up to Day 45
  Descriptively summarize at baseline and post-immunotherapy treatments.

SECONDARY OUTCOMES:
change of SUVpeak | Up to Day 45
  Descriptively summarize the percent change from baseline to post-immunotherapy treatments.
change of SUVmean | Up to Day 45
  Descriptively summarize the percent change from baseline to post-immunotherapy treatments.
change of SUVmax | Up to Day 45
  Descriptively summarize the percent change from baseline to post-immunotherapy treatments.

OTHER OUTCOMES:
change of SUVpeak by PET response | Up to Day 45
  Descriptively summarize the percent change from baseline to post-immunotherapy by PET response
change of SUVmean by PET response | Up to Day 45
  Descriptively summarize the percent change from baseline to post-immunotherapy by PET response
change of SUVmax by PET response | Up to Day 45
  Descriptively summarize the percent change from baseline to post-immunotherapy by PET response

CONTACTS AND LOCATIONS:
Overall Officials: Nerissa T Viola, PhD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No